CLINICAL TRIAL: NCT07221903
Title: The Lateral, Anterior, Medial (LAM) Femoral Cutaneous Block: A Case Series Harborview Medical Center, Seattle, WA
Acronym: LAM
Status: Recruiting | Type: Observational
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Dorothy Wang, Acting Assistant Professor, Department of Anesthesiology and Pain Medicine, University of Washington
Other Study IDs: STUDY00023101
Record Dates: First submitted 2025-10-24; First posted 2025-10-28 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-10

CONDITIONS: Regional Anesthesia; Burn; Skin Grafting
MeSH Terms: conditions — Burns

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Skin donor sites in patients undergoing split-thickness skin grafting surgeries can be very painful postoperatively. This site is most often the anterolateral thigh, the pain at which location can traditionally be covered by a fascia iliaca nerve block, although that comes with the disadvantage of losing motor functions in the femoral nerve distribution. The LAM nerve block, which is relatively new, aims to provide analgesia in the distribution of the lateral and anterior femoral cutaneous nerves. In short, this nerve block would decrease the sensation of the anterolateral thigh area without affecting the motor function of the leg. Investigators aim to study the consistency and coverage size of sensation changes by mapping out the area after the block in each patient.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years or older
2. Scheduled surgery for STSG w/ donor site coming from thigh
3. Care team requests LAM nerve block
4. Anticipated postop pain in the cutaneous areas of anterior and lateral thigh

   Exclusion Criteria:
5. Inability to communicate sensation or motor changes in their body
6. Preexisting sensory or motor deficits in the femoral nerve distribution
7. Contraindication to the medication used or a peripheral nerve block, such as allergy to amide local anesthetics, severe liver dysfunction, injection site infection etc
8. Pregnancy
9. Prisoners
10. Non-English Speaking/reading
11. Surgeries with anticipated or actual duration of 6 hours or longer
12. TBSA 20% or greater
13. Severe distracting injuries/polytrauma (e.g., large or significant bone fractures)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 18 years or older who are undergoing skin grafting surgeries
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2025-10-22 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Area of sensory change after nerve block | 20 min after nerve block placement

CONTACTS AND LOCATIONS:
Overall Officials: Dorothy Wang, MD, MHA, Principal Investigator — University of Washington
Locations (1):
- Harborview Medical Center, Seattle, Washington, United States